CLINICAL TRIAL: NCT00983710
Title: Prostate Cancer Symptom Management for Low Literacy Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Latini, Associate Professor of Urology, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MRSGT-06-083-01-CPPB; NCT00903123 (obsolete NCT alias); NCT00903487 (obsolete NCT alias)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: prostate neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive a new patient education program designed to help men manage side-effects related to treatment for localized prostate cancer. The intervention will be targeted to low health literacy men.
  Interventions: Behavioral: PC-PEP - Prostate Cancer Patient Education Program
- 2 (Active Comparator): Usual care, including a booklet on coping with localized prostate cancer. After the 6-month primary outcome data are collected, control group men will be offered the opportunity to cross-over and receive the new educational intervention.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PC-PEP - Prostate Cancer Patient Education Program — Men in the intervention group will receive a new patient education intervention to help them manage side-effects related to treatment for localized prostate cancer. The intervention will be delivered by phone and by mail and is targeted to me with low health literacy. The intervention consists of written materials, audio materials, and telephone-based problem-solving education.
  Arms: 1
Behavioral: Usual care — Booklet on coping with localized prostate cancer
  Arms: 2

SUMMARY:
This study will compare a newly-developed patient education program to help men with localized prostate cancer manage treatment-related side-effects versus usual care. The new intervention will be developed for men with lower health literacy. That means that the education materials will be developed for sixth grade reading level or lower. The materials will include lots of examples and illustrations to make it easier for people understand the information.

DETAILED DESCRIPTION:
Prostate cancer has recently surpassed lung cancer to become the most common cancer of American men. The estimated number of new prostate cancer cases in 2005 is expected to be 232,090, up from 198,000 in 2002. Prostate cancer represents 29% of all new cancer diagnoses in men and is comparable to the incidence of breast cancer in women. Prostate cancer continues to disproportionately affect minority men. For patients with early, localized prostate cancer, there are a number of treatment options, including surgical removal of the prostate, radiation therapy (external beam or implantation of radioactive "seeds"), hormonal therapy, cryoablation, or expectant monitoring ("watchful waiting"). Most of these currently available treatments for localized prostate cancer carry the risk of a number of iatrogenic symptoms, including urinary incontinence, ED, and others that vary depending on the treatment received.

The need for symptom management education is greater for men with lower health literacy. Health literacy - "the ability to which individuals have the capacity to obtain, process, and understand health information services needed to make appropriate health decisions" - has been shown to be strongly related to health status and health outcomes. Persons with lower health literacy skills are significantly less likely to take preventive actions to improve their health. Health literacy is a particular concern for men with prostate cancer because African-American men, a group with a significantly higher prevalence of prostate cancer, are over-represented among lower literacy men with prostate cancer.3 The study proposed here will develop and evaluate in a randomized controlled trial (RCT) an empirically-derived symptom management intervention for lower literacy men with prostate cancer. The intervention will be based on a biopsychosocial model of prostate cancer symptom management developed from the more general the UCSF Symptom Management Model (SMM) and Bandura's Self-Efficacy Theory.

The efficacy of the intervention will be evaluated with 200 men with localized prostate cancer randomized to receive either the new tailored symptom management program or usual care. Participants in both the intervention and control groups will receive a booklet on coping with cancer available to all patients treated at the UCSF Comprehensive Cancer Center. Intervention group participants also will receive a new symptom management intervention tailored to their individual symptom profile. Both groups will be followed for 6 months after enrollment, with assessments at enrollment and 5 additional timepoints.

The proposed research project includes the following specific aims:

1. Conduct an RCT to evaluate a tailored symptom management intervention targeted to lower literacy men with localized prostate cancer.

   The investigators hypothesize men who receive the tailored symptom management intervention (N=100) will report significantly less symptom distress at the 6-month follow-up than men in the control condition (N=100). Symptom distress will be measured by the Expanded Prostate Cancer Index Composite (EPIC) Urinary Bother and Sexual Bother sub-scales. The intervention and control groups will be stratified by literacy level and type of prostate cancer treatment.
2. Complete a planned training experience that will include courses in responsible conduct of research, symptom management, cancer care, cancer prevention, cancer epidemiology, clinical research with diverse communities, and longitudinal analysis methods that will provide the knowledge and skills necessary to successfully conduct the RCT.
3. Assemble a group of key personnel with expertise necessary to guide the training experience and RCT. The primary mentor will be Leslie Schover, PhD, an expert in cancer symptom management. Other key personnel will include Stephen J. Lepore, PhD, Principal Investigator of a previous prostate cancer psychosocial intervention study; Brian J. Miles, MD, an expert in prostate cancer treatment; and Robert Morgan, PhD, a senior methodologist.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. 18 years or older, with biopsy-proven prostate cancer
3. Diagnosed with localized disease in the preceding 2 years
4. Have a telephone at the time of enrollment
5. Have an address where they can receive intervention materials by mail
6. Able to speak and understand English
7. Treated with radiation, surgery, or hormonal therapy
8. Receive prostate cancer treatment and follow-up at the Michael E DeBakey VA Medical Center in Houston, TX

Exclusion Criteria:

1. Younger than 18
2. Female
3. Diagnosis of advanced prostate cancer
4. No treatment for prostate cancer
5. Diagnosed with localized disease more than 2 years before trial enrollment
6. Unable to speak and understand English
7. Unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Sexual Bother score from Expanded Prostate Cancer Index Urinary Bother score from Expanded Prostate Cancer Index | Six months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: David M Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States